CLINICAL TRIAL: NCT07377942
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial Assessing Gut Health and Immunomodulatory Effects of Bacillus Subtilis-based Product in Healthy Adults
Brief Title: To Evaluate the Effect of Bacillus Subtilis Based Product in Gut Health and Immunomodulatory Effect in Healthy Adults.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bioagile Therapeutics Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BSP-25-072
Record Dates: First submitted 2026-01-05; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants Study
Keywords: Gut Health and Immunomodulatory effect
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Bacillus subtilis
  Interventions: Dietary Supplement: Probiotics (Bacillus Subtilis)
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics (Bacillus Subtilis) — Experimental
  Arms: Probiotics
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to Assess Gut Health and Immunomodulatory Effects of Bacillus Subtilis based product in Healthy Adults The main question[s] it aims to answer are to assess the effects of Bacillus Subtilis on gut health in healthy adults by measuring changes in fecal calprotectin levels as a marker of intestinal inflammation, in comparison between the intervention and placebo group.

To assess the immunomodulatory effects of Bacillus-Subtilis by measuring changes in inflammatory and immune response markers, in comparison between the intervention and placebo group To confirm the safety and tolerability of the study product Bacillus Subtilis in the healthy study population during the intended use, with safety assessments conducted across both the intervention and placebo groups.

The primary and secondary outcomes are:

Primary Efficacy Outcome:

* Change in fecal calprotectin levels from baseline to the end of the study, comparing the intervention and placebo groups.
* Changes in immunological markers (IgA, IgG, IgM) between baseline and study completion, comparing the intervention and placebo groups.

Secondary Efficacy Outcome:

• Improvement in the patient related overall relief, assessed using Gut Health Status Questionnaire (GHSQ) and Immune status questionnaire (ISQ) score with comparative analysis between the two groups.

Participants will be asked to take the probiotics twice daily morning and evening after meals and record it in the subject diary.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18 and 50 years.
2. Female participants are either not of childbearing potential, or females of childbearing potential agree to use a medically approved method of birth control and have a negative urine pregnancy test result.
3. In good general health, as determined by medical history, laboratory analysis, and physical examination performed by the study physician.
4. Willing to provide fecal samples as per the study requirements.
5. Willing to participate voluntarily and provide written informed consent.

Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Subjects who are taking Antibiotic treatment.
3. Subjects suffering from Gastrointestinal disease.
4. Subjects suffering from Diabetes.
5. Subjects suffering from Chronic/iatrogenic Immunodeficiency.
6. Subjects suffering from Abnormal blood pressure.
7. Subjects who are allergic to ingredients of the study Product.
8. Subjects who are Smoker or alcoholic.
9. Subjects who have participated prior in conflicting clinical trial or have participated in the trial over the last 3months.
10. Women who are pregnant, breastfeeding, or planning to become pregnant.
11. Daily use of supplements that contain probiotics or prebiotics within 30 days prior to screening or during study.
12. Subjects with medical conditions affecting immune status (e.g., rheumatoid arthritis, heart failure, hepatitis C, HIV) or taking medications that may impact the immune system, such as antibiotics, antimicrobials, or probiotic sachets.
13. Any surgical treatment within the previous three months or planned during the study.
14. Any subject, in the principal investigator's opinion, not considered suitable for enrolment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
• Change in fecal calprotectin levels from baseline to the end of the study. | Baseline to Week 8 (or end of study)
  Fecal calprotectin concentration (µg/g) will be measured at baseline and at the end of the study. The change from baseline will be analyzed.

SECONDARY OUTCOMES:
Change in Gut Health Status Questionnaire (GHSQ) Total Score from Baseline to End of Study | Baseline to Week 8 (End of Study)
  The Gut Health Status Questionnaire (GHSQ) total score will be assessed at baseline and at the end of the study. The change from baseline will be analyzed.
Change in Serum Immunoglobulin A (IgA) Concentration from Baseline to End of Study | Baseline to Week 8 (or end of study)
  Serum IgA concentration (mg/dL) will be measured at baseline and at study completion, and the change from baseline will be assessed.
Change in Serum Immunoglobulin G (IgG) Concentration from Baseline to End of Study | Baseline to Week 8 (or end of study)
  Serum IgG concentration (mg/dL) will be measured at baseline and at study completion, and the change from baseline will be assessed.
Change in Serum Immunoglobulin M (IgM) Concentration from Baseline to End of Study | Baseline to Week 8 (or end of study)
  Serum IgM concentration (mg/dL) will be measured at baseline and at study completion, and the change from baseline will be assessed.
Change in Immune Status Questionnaire (ISQ) Total Score from Baseline to End of Study | Baseline to Week 8 (End of Study)
  The Immune Status Questionnaire (ISQ) total score will be assessed at baseline and at the end of the study. The change from baseline will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Parag Saudagar, Study Director — S K Biobiz Private Limited
Locations (1):
- Advanced Gastro Care, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No